CLINICAL TRIAL: NCT05392504
Title: Effects of Core Stabilization Exercises Versus Schroth's Program on Posture and Quality of Life in Females With Idiopathic Scoliosis.
Brief Title: Effects of Core Stabilization Exercises vs. Schroth's Program on Posture and Quality of Life in Females With Scoliosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0519
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Scoliosis Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability exercise (Experimental): The core stability training consist of three phases. The first and second phases each will last for three weeks in total, and the third phase will take place in four weeks. Each training session will begin with 10 minutes of warm-up exercises and finish with 10 minutes of cool-down exercises; both warm-up and cool-down exercises includes breathing and stretching exercises. The number of repetitions will be adjusted according to the participant's exercise tolerance.
  During the first week of each phase, the number of repetitions of each exercise will be 7-10, and this will progress to 10-15 based on the patient's physical tolerance.
  Interventions: Other: Core stability exercise
- Scroth's program (Active Comparator): The Schroth program include exercises for rotational breathing, spinal elongation, de-flexion, stretching, de-rotation, and strengthening, and these exercises are performed to improve the curvature, muscle strength, and endurance of postural muscles. During the Schroth exercises, rice bags, foam blocks, a stool, and long sticks will be used to adjust the posture and give passive support. The intensity of the Schroth exercises will gradually increased depending on the patient's improvement in exercise performance by decreasing the amount or degree of passive support, changing the patient's position, and adjusting the sets and repetitions of exercises
  Interventions: Other: Scroth's Program

INTERVENTIONS:
Other: Core stability exercise — The core stability training consist of three phases
  Arms: Core stability exercise
Other: Scroth's Program — The Schroth program include exercises for rotational breathing, spinal elongation, deflexion, stretching, de-rotation, and strengthening
  Arms: Scroth's program

SUMMARY:
The objective of this study is to compare the effects of core stabilization exercises versus schroth's program on posture and quality of life in females with idiopathic scoliosis

DETAILED DESCRIPTION:
Scoliosis is a 3 dimension condition that effects most of our population specifically females. It is not only a bend in your spine but according to new research, its also twisting it. The curvature effects the effected individual physical and the social anxiety due to appearance and a continues state of lethargy effects their quality of life immensely. The posture is poorly effected along with a visual appearance. Often someone with scoliosis might find good posture difficult. Often someone with scoliosis will lean forwards and to the side either slightly or a lot. They will often try to avoid doing this, which can lead to slightly bent knees and the pelvis tilting backwards. Scoliosis is often defined as spinal curvature in the "coronal" (frontal) plane. While the degree of curvature is measured on the coronal plane, scoliosis is actually a more complex, three-dimensional problem which involves all 3 planes. It is defined by the Cobb's angle of spine curvature in the coronal plane and is often accompanied by vertebral rotation in the transverse plane and hypokyphosis in the sagittal plane. These abnormalities in the spine, costal-vertebral joints, and the rib cage produce a 'convex' and 'concave' hemithorax.

Only females having idiopathic scoliosis with cob's angle 10°-26° with age ranging between 19-30 are included and any subjects with surgical interventions are excluded.

Population will be divided in to two groups. One group will perform scroth exercises for 4 weeks and the other group will perform core straightening exercises for 4 weeks each. Once the time period is complete, the posture will be measured using pelvic and shoulder goniometers to check the level of tilt and for quality of lifestyle, we will be using quality of life (Scoliosis Research Society-22 questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Females only
* Positive Forward bend test (FBT)
* Idiopathic scoliosis
* Cob's angle 10°-26°
* Age group ranged between 19-30 yrs.
* Normal BMI (18.5-24.9 kg/m2)
* Chronic Scoliosis patients
* Riser Sign 4-5

Exclusion Criteria:

* Subjects with any surgical intervention for scoliosis
* Pregnant women
* Subjects with any serious health condition

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Scoliosis Research Society-22 questionnaire | 4 week
  It is a standardized questionnaire designed by scoliosis research society to measure the quality of life in scoliosis patients. Each item is scored from 1 (worst) to 5 (best). Each domain has a total sum score ranging from 5 to 25, except for satisfaction, which ranges from 2 to 10. The sum of the first 4 domains gives a maximum subtotal of 100, and when the satisfaction domain is included, the maximum total is 110.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, Ms, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - New canal medical center, Lahore, Punjab Province
  - Pakistan Society for the Rehabilitation of the Disabled, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dela Merced P, Vazquez Colon C, Mirzada A, Oke A, Gal Z, Cheng J, Oetgen MM, Martin B, Pestieau SR, Cronin JA. Association between implementation of a coordinated care pathway in idiopathic scoliosis patients and a reduction in perioperative outcome disparities. Paediatr Anaesth. 2022 Apr;32(4):556-562. doi: 10.1111/pan.14330. Epub 2021 Dec 10. PMID 34758176
- [Background] Mesiti BL. Scoliosis: An Overview. Radiol Technol. 2021 Sep;93(1):55-72. PMID 34588279
- [Background] Janicki JA, Alman B. Scoliosis: Review of diagnosis and treatment. Paediatr Child Health. 2007 Nov;12(9):771-6. doi: 10.1093/pch/12.9.771. PMID 19030463
- [Background] Sun Y, Xing Y, Zhao Z, Meng X, Xu G, Hai Y. Comparison of manual versus automated measurement of Cobb angle in idiopathic scoliosis based on a deep learning keypoint detection technology. Eur Spine J. 2022 Aug;31(8):1969-1978. doi: 10.1007/s00586-021-07025-6. Epub 2021 Oct 30. PMID 34716822
- [Background] Ren J, Liu X, Chen F, Jing X, Cui X. Association Between Vertebral Rotatory Subluxation and the Apical Vertebra in Degenerative Lumbar Scoliosis. World Neurosurg. 2021 Oct;154:e627-e632. doi: 10.1016/j.wneu.2021.07.101. Epub 2021 Jul 28. PMID 34329750
- [Background] Liang JQ, Qiu GX, Shen JX, Lee CI, Wang YP, Zhang JG, Zhao H. A retrospective study of echocardiographic cardiac function and structure in adolescents with congenital scoliosis. Chin Med J (Engl). 2009 Apr 20;122(8):906-10. PMID 19493412
- [Background] Grunwald ATD, Roy S, Alves-Pinto A, Lampe R. Assessment of adolescent idiopathic scoliosis from body scanner image by finite element simulations. PLoS One. 2021 Feb 10;16(2):e0243736. doi: 10.1371/journal.pone.0243736. eCollection 2021. PMID 33566808
- [Background] Zhou Z, Liu F, Li R, Chen X. The effects of exercise therapy on adolescent idiopathic scoliosis: An overview of systematic reviews and meta-analyses. Complement Ther Med. 2021 May;58:102697. doi: 10.1016/j.ctim.2021.102697. Epub 2021 Feb 23. PMID 33636298
- [Background] Yan B, Lu X, Qiu Q, Nie G, Huang Y. Association Between Incorrect Posture and Adolescent Idiopathic Scoliosis Among Chinese Adolescents: Findings From a Large-Scale Population-Based Study. Front Pediatr. 2020 Sep 15;8:548. doi: 10.3389/fped.2020.00548. eCollection 2020. PMID 33042909
- [Background] Ko JY, Suh JH, Kim H, Ryu JS. Proposal of a new exercise protocol for idiopathic scoliosis: A preliminary study. Medicine (Baltimore). 2018 Dec;97(49):e13336. doi: 10.1097/MD.0000000000013336. PMID 30544395
- [Background] Makino T, Kaito T, Kashii M, Iwasaki M, Yoshikawa H. Low back pain and patient-reported QOL outcomes in patients with adolescent idiopathic scoliosis without corrective surgery. Springerplus. 2015 Aug 7;4:397. doi: 10.1186/s40064-015-1189-y. eCollection 2015. PMID 26261755
- [Background] Aulisa AG, Guzzanti V, Perisano C, Marzetti E, Specchia A, Galli M, Giordano M, Aulisa L. Determination of quality of life in adolescents with idiopathic scoliosis subjected to conservative treatment. Scoliosis. 2010 Sep 28;5:21. doi: 10.1186/1748-7161-5-21. PMID 20920196
- [Background] Gur G, Ayhan C, Yakut Y. The effectiveness of core stabilization exercise in adolescent idiopathic scoliosis: A randomized controlled trial. Prosthet Orthot Int. 2017 Jun;41(3):303-310. doi: 10.1177/0309364616664151. Epub 2016 Sep 13. PMID 27625122
- [Background] Radwan NL, Ibrahim MM, Mahmoud WS. Comparison of two periods of Schroth exercises for improving postural stability indices and Cobb angle in adolescent idiopathic scoliosis. J Back Musculoskelet Rehabil. 2022;35(3):573-582. doi: 10.3233/BMR-200342. PMID 34602457
- [Background] Beardsley C, Egerton T, Skinner B. Test-re-test reliability and inter-rater reliability of a digital pelvic inclinometer in young, healthy males and females. PeerJ. 2016 Mar 31;4:e1881. doi: 10.7717/peerj.1881. eCollection 2016. PMID 27069812
- [Background] Korbel K, Kinel E, Janusz P, Kozinoga M, Czaprowski D, Kotwicki T. The measurement of health-related quality of life of patients with idiopathic scoliosis - comparison of ISYQOL versus SRS-22 questionnaire. Stud Health Technol Inform. 2021 Jun 28;280:323. doi: 10.3233/SHTI210529. No abstract available. PMID 34190141